CLINICAL TRIAL: NCT02948465
Title: Impact of Neutrophil Extracellular Traps (NET) on Thrombolysis in Acute Phase of Cerebral Ischemia
Acronym: THINK
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/37
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Cerebral Infarct
Keywords: Neutrophil Extracellular Traps
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cerebral infarcts represent a major cause of morbidity/mortality in spite of therapeutics for a premature recanalisation (intravenous recombinant tissue plasminogen activator (rt-PA) and thrombectomy). Thrombolysis failure by the administration of rt-PA is frequent, in particular in proximal occlusion. Experimental studies suggest that neutrophils could play an important role in the thrombus development via the organization of a network (NET) within the thrombus. Targeting this network of NET could, in addition to the fibrinolysis, increase the rate of recanalisation and thus improve the neurological prognostic after a cerebral infarct.

The aim of the research is to Study of the biochemical and histological composition of the stemming thrombi of cerebral thrombectomies with in vitro analysis of the sensibility in the thrombolysis induced by rt-PA +/- Desoxyribonuclease I (DNase I).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18
* Having a cerebral infarct consecutive to a wide calibre arterial occlusion
* taken care for mechanical thrombectomy

Exclusion Criteria:

* Patient benefiting from a legal protective measure
* Pregnant or breast-feeding woman
* Opposition of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cerebral infact after wide calibre arterial occlusion
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2016-12-10 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient between biochemical and histological composition of the thrombus and the sensibility in the in vitro fibrinolysis and the origin of the thrombus. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Arturo CONSOLI, MD, Principal Investigator — Hopital Foch; Bertrand LAPERGUE, MD, Study Chair — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No